CLINICAL TRIAL: NCT00051311
Title: A Pilot Study of EPOCH-F/R Induction Chemotherapy and Reduced-Intensity, HLA-Matched, Related Allogeneic Hematopoietic Stem Cell Transplantation, With Cyclosporine & Methotrexate GVHD Prophylaxis for Refractory or Relapsed Hematologic Malignancies
Brief Title: Modified Stem Cell Transplant Procedure to Treat Patients With Blood and Immune System Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ronald Gress, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 030077; 03-C-0077; NCT00055744 (obsolete NCT alias)
Record Dates: First submitted 2003-01-08; First posted 2003-01-08 (Estimated); Results first posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-08

CONDITIONS: Hematologic Neoplasms
Keywords: Lymphoma; Leukemia; Hodgkin's Disease; Multiple Myeloma; Immunotherapy
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma; Leukemia; Hodgkin Disease; Multiple Myeloma | interventions — Stem Cell Transplantation; fludarabine; fludarabine phosphate; Cyclophosphamide; Etoposide; Doxorubicin; liposomal doxorubicin; Vincristine; Prednisone; Methotrexate; Cyclosporine; Blood Component Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Donor (Other): Donors will undergo apheresis to collect stem cells for a stem cell transplant for the recipient.
  Interventions: Procedure: Apheresis
- Recipient (Experimental): Recipients will receive induction chemotherapy (one cycle is 5 days on drug therapy followed by a 16 day rest period). Prior to the transplant procedure, recipients will receive conditioning therapy followed by the infusion of donor stem cells.
  Interventions: Procedure: Stem cell transplantation; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Etoposide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Methotrexate; Drug: Cyclosporine

INTERVENTIONS:
Procedure: Stem cell transplantation — Recipients will receive donor stem cells 3 days after conditioning therapy is completed.
  Other Names: hematopoietic stem cell transplant (HSCT)
  Arms: Recipient
Drug: Fludarabine — Recipients will receive induction therapy with fludarabine, cyclophosphamide, etoposide, doxorubicin, vincristine, and prednisone. One cycle is 5 days on drug therapy followed by a 16 day rest period.
  Other Names: Fludara
  Arms: Recipient
Drug: Cyclophosphamide — Recipients will receive induction therapy with fludarabine, cyclophosphamide, etoposide, doxorubicin, vincristine, and prednisone. One cycle is 5 days on drug therapy followed by a 16 day rest period.
  Other Names: Cytoxan
  Arms: Recipient
Drug: Etoposide — Recipients will receive induction therapy with fludarabine, cyclophosphamide, etoposide, doxorubicin, vincristine, and prednisone. One cycle is 5 days on drug therapy followed by a 16 day rest period.
  Other Names: Toposar
  Arms: Recipient
Drug: Doxorubicin — Recipients will receive induction therapy with fludarabine, cyclophosphamide, etoposide, doxorubicin, vincristine, and prednisone. One cycle is 5 days on drug therapy followed by a 16 day rest period.
  Other Names: Doxil
  Arms: Recipient
Drug: Vincristine — Recipients will receive induction therapy with fludarabine, cyclophosphamide, etoposide, doxorubicin, vincristine, and prednisone. One cycle is 5 days on drug therapy followed by a 16 day rest period.
  Other Names: Oncovin
  Arms: Recipient
Drug: Prednisone — Recipients will receive induction therapy with fludarabine, cyclophosphamide, etoposide, doxorubicin, vincristine, and prednisone. One cycle is 5 days on drug therapy followed by a 16 day rest period.
  Other Names: Deltasone
  Arms: Recipient
Drug: Methotrexate — Recipients will receive 4 doses of methotrexate by vein after the transplant to help prevent graft-versus-host disease (GVHD)..
  Other Names: Rasuvo
  Arms: Recipient
Drug: Cyclosporine — Recipients will receive cyclosporine by vein or by mouth for about 6 months after the transplant to help prevent graft-versus-host disease (GVHD).
  Other Names: Neoral
  Arms: Recipient
Procedure: Apheresis — Donors will undergo apheresis to collect stem cells for a stem cell transplant for the recipient.
  Other Names: extracorporeal therapy
  Arms: Donor

SUMMARY:
This study will investigate the safety and effectiveness of a modified stem cell transplant procedure for treating cancers of the blood and immune system. Patients with cancers and pre-cancerous conditions originating in blood or immune system cells can sometimes benefit greatly from, and even be cured by, transplants of stem cells (cells produced by the bone marrow that mature into blood cells). In addition to producing new bone marrow and restoring normal blood production and immunity, the donated cells fight any residual tumor cells that might have remained in the body, in what is called a graft-versus-tumor effect.

However, severe problems, and sometimes death, may follow these transplants as a result of the high-dose chemotherapy and radiation that accompany the procedure. Also, donated immune system cells called T cells sometimes attack healthy tissues in a reaction called graft-versus-host-disease (GVHD), damaging organs such as the liver, intestines and skin. This study will use the following strategies to try to reduce these risks:

* induction chemotherapy to reduce patient's immunity in an attempt to prevent rejection of the donated stem cells;
* reduced-intensity conditioning chemotherapy that is easier for the body to tolerate and involves a shorter period of complete immune suppression;
* donation of immune cells called T helper type 2 (Th2) cells instead of T cells to try to reduce the risk of serious GVHD;
* treatment with methotrexate and cyclosporine to try to reduce the risk of serious GVHD.

Patients between 12 and 75 years of age with non-Hodgkin's lymphoma, Hodgkin's lymphoma, multiple myeloma, chronic lymphocytic leukemia, chronic myelogenous leukemia, acute myelogenous leukemia, acute lymphocytic leukemia, myelodysplasia, idiopathic myelofibrosis, polycythemia vera, or chronic myelomonocytic leukemia may be eligible for this study. Candidates will have a medical history, physical and dental examinations, blood and urine tests (including a blood test for genetic match with the donor), lung and heart function tests, and X-ray studies. A bone marrow biopsy may be done to evaluate disease status. Patients with lymphoma may have a nuclear medicine test called a positron emission tomography (PET) scan.

Participants will have a central venous line (large plastic tube) placed into a major vein. This tube can stay in the body and be used during the entire treatment period to deliver the donated stem cells and give medications, including chemotherapy and other drugs, antibiotics and blood transfusions, and to withdraw blood samples. Treatment will start with induction chemotherapy, which will include the drugs fludarabine, cyclophosphamide, etoposide, doxorubicin, vincristine, and prednisone. Some patients may also receive an antibody called rituximab. Patients will receive one to three cycles of this treatment, depending on their response to the drugs. (One cycle consists of 5 days on drug therapy followed by a 16-day rest period.) Several days before the transplant procedure, patients will start conditioning chemotherapy with cyclophosphamide and fludarabine. Three days after the conditioning therapy is completed, the stem cells will be infused. To help prevent GVHD, patients will take four doses of methotrexate (by vein) shortly after the transplant, and cyclosporine (by mouth or by vein) for about 6 months after the transplant.

The average hospital stay for stem cell transplantation is 3 to 4 weeks. After discharge, patients will return for frequent follow-up visits for 3 months. Monthly visits will be scheduled for the next 3 months, then every 3 months for the next 18 months, and less frequently for a total of at least 5 years post-transplant. These visits will include bone marrow aspirates and biopsies, blood draws, and other tests to monitor disease status.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (HSCT) is potentially curative for refractory hematologic malignancies, but its application has been limited historically by morbidity and mortality from conventional transplant preparative regimens and graft-versus-host disease (GVHD). Donor T cells mediate GVHD and also help to eradicate malignancies through an immune-dependent graft-versus-tumor effect. Efforts to decrease preparative regimen toxicity have led to reduced-intensity or 'nonmyeloablative' regimens, facilitating the study of allogeneic HSCT in a broader population. As a promising strategy for reducing GVHD, donor T helper type 2 (Th2) cells were shown to abrogate T helper type 1 (Th1)-mediated GVHD without impairing engraftment in murine models of allogeneic HSCT. These findings led to a phase I/II clinical study of donor Th2 cells for the prevention of GVHD during reduced-intensity allogeneic HSCT (CC 99-C-0143); preliminary results suggest that a randomized trial will be necessary to evaluate donor Th2 cells further.

In CC 99-C-0143, a novel induction chemotherapy regimen, etoposide phosphate, prednisone, vincristine sulfate, cyclophosphamide, and doxorubicin hydrochloride (EPOCH)-Fludarabine (EPOCH-F), was well tolerated and effective for sequential host immune depletion. However, a significant proportion of patients failed to achieve satisfactory disease control before transplant, providing a basis for intensifying this induction regimen. Furthermore, the initial 20 patients treated on this study experienced relatively high rates of acute GVHD and considerable morbidity associated with cyclosporine monotherapy for GVHD prevention, indicating that future studies should use more aggressive prophylaxis. These observations warrant modifying our approach to allogeneic HSCT before undertaking a randomized study of donor Th2 cells.

We now propose a pilot study of human leukocyte antigens (HLA)-matched, related, reduced-intensity allogeneic HSCT in refractory hematologic malignancies, using an intensified etoposide, vincristine, doxorubicin, prednisone, cyclophosphamide and fludarabine (EPOCH-F) induction chemotherapy regimen with rituximab added for patients with cluster of differentiation 20 (CD20)+ malignancies fludarabine, etoposide, prednisone, vincristine, cyclophosphamide, and doxorubicin plus with or without rituximab (DA-EPOCH-F/R). This regimen will be evaluated for toxicity and disease control before transplantation. GVHD prophylaxis will consist of a standard dual-agent regimen, cyclosporine/methotrexate; the impact of this change on hematopoietic recovery, donor/recipient chimerism, and the incidence of acute GVHD will be assessed.

Immune reconstitution following allogeneic HSCT is an important research interest among Experimental Transplantation and Immunology Branch Investigators. Current evidence suggests a critical role for interleukin-7 (IL-7) in cluster of differentiation 4 (CD4)+ T cell homeostasis, and interleukin-15 (IL-15) appears crucial to cluster of differentiation 8 (CD8)+ T cell and NK cell homeostasis. The relationships between these cytokines and lymphocyte subpopulations have not been studied in the setting of allogeneic HSCT; such analysis may enhance our understanding of engraftment kinetics, graft-versus-host disease, and immune reconstitution. We will correlate serum IL-7 and IL-15 levels with changes in circulating T-cell and natural killer (NK)-cell subpopulations during EPOCH-F/R induction chemotherapy, after transplantation, and with the development of GVHD.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion Criteria Patient (Recipient):

Patients with hematologic malignancies, myelodysplasia, or myeloproliferative disorders, as summarized below:

Disease: Chronic Lymphocytic Leukemia; Disease Status: (a) Relapse post-fludarabine, (b) Non-Complete Remission (CR) after salvage regimen; Age: 18 to 75.

Disease: Hodgkin's and Non-Hodgkin's Lymphoma (all types, including Mantle Cell Lymphoma); Disease Status: (a) Primary treatment failure, (b) Relapse after autologous stem cell transplant (SCT), (c) Hepatosplenic gamma/delta T cell lymphoma; Age: 18 to 75.

Disease: Multiple Myeloma; Disease Status: (a) Primary treatment failure, (b) Relapse after autologous SCT, (c) Non-CR after salvage regimen; Age: 18 to 75.

Disease: Acute Myelogenous Leukemia; Disease Status: (a) In Complete Remission #1, with high-risk cytogenetics [abnormalities other than t(8;21), t(15;17), or inv(16)], (b) In Complete Remission #2 or greater; Age: 18 to 75.

Disease: Acute Lymphocytic Leukemia; Disease Status: (a) In Complete Remission #1, with high-risk cytogenetics [t(9;22) or bcr-abl rearrangement; t(4;11), 1(1;19), t(8;14)], (b) In Complete Remission #2 or greater; Age: 18 to 75.

Disease: Myelodysplastic Syndrome; Disease Status: (a) refractory anemia with excess blasts (RAEB), (b) refractory anemia with excess blasts in transformation (RAEB-T) (if blasts are less than 10% in marrow and blood after induction chemotherapy); Age: 18 to 75.

Disease: Myeloproliferative disorders; Disease Status: (a) Idiopathic myelofibrosis, (b) Polycythemia vera, (c) Essential thrombocytosis, (d) Chronic myelomonocytic leukemia; Age: 18 to 75.

Disease: Chronic Myelogenous Leukemia (CML); Disease Status: (a) Chronic phase CML, (b) Accelerated phase CML; Age 50 to 75; (c) Not eligible for myeloablative allogeneic HSCT; Age: 18 to 50.

Patients 18-75 years of age. Patients older than 75 years of age will be considered on an individual basis.

Consenting first degree relative matched at 6/6 human leukocyte antigen (HLA) antigens (A, B, and DR).

Patient or legal guardian must be able to give informed consent.

All previous therapy must be completed at least 2 weeks prior to study entry, and any grade 3 or 4 non-hematologic toxicity of previous therapy must be resolved to grade 2 or less, unless specified elsewhere.

Eastern Cooperative Oncology Group (ECOG) performance status equal to 0 or 1.

Life expectancy of at least 3 months.

Patients with acute leukemia must be in hematologic remission, defined as less than 5% blasts present in blood or bone marrow.

Left ventricular ejection fraction greater than 45% by either multi-gated acquisition (MUGA) scan or 2-D echo, obtained within 28 days of enrollment. The cumulative dose of doxorubicin received by patients will not be considered, as the cardiac ejection fraction appears to indicate the safe cumulative doxorubicin dose in the setting of etoposide phosphate, prednisone, vincristine, cyclophosphamide, and doxorubicin hydrochloride (EPOCH)-based chemotherapy.

Diffusing capacity for carbon monoxide (DLCO) greater than 50% of the expected value when correlated for hemoglobin (Hb), obtained within 28 days of enrollment.

Creatinine less than or equal to 1.5 mg/dl and creatinine clearance greater than or equal to 50 ml/min/1.73 m(2).

Serum total bilirubin less than 2.5 mg/dl, and serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) values less than or equal to 2.5 times the upper limit of normal. Values above these levels may be accepted, at the discretion of the principal investigator (PI) or study chairman, if such elevations are thought to be due to liver involvement by malignancy. If these values do not normalize during induction chemotherapy, such patients will not be eligible for the transplant phase of the protocol, and will thus be taken off study.

Minimum absolute neutrophil count of 1,000 cells/microliter and minimum platelet count (without transfusion) of 20,000/mm(3).

Inclusion Criteria Donor:

First-degree relative with genotypic identity at 6/6 HLA loci (HLA-A, B and DR).

Ability to give informed consent. For donors under 18 years of age, the donor must complete an assent form, and the donors legal guardian must complete an informed consent form.

Age 12-75 years. As the potential cerebrovascular and cardiac complications may potentially increase with age, age 75 has been chosen arbitrarily as the upper age limit. However, if it is determined after initial accrual of patients in this upper age range that this procedure is relatively safe, the age range may be extended.

Adequate venous access for peripheral apheresis, or consent to use a temporary central venous catheter for apheresis.

Donors must be human immunodeficiency virus (HIV) negative, hepatitis B surface antigen negative, and hepatitis C antibody negative. This is to prevent the possible transmission of these infections to the recipient.

A donor who is lactating must substitute formula feeding for her infant during the period of cytokine administration. Filgrastim may be secreted in human milk, although its bioavailability from this source is not known. Limited clinical data suggest that short-term administration of filgrastim or sargramostim to neonates is not associated with adverse outcomes.

EXCLUSION CRITERIA:

Exclusion Criteria Patient:

Active infection that is not responding to antimicrobial therapy.

Active central nervous system (CNS) involvement by malignancy.

HIV infection. There is theoretical concern that the degree of immune suppression associated with the treatment may result in progression of HIV infection.

Chronic active hepatitis B. Patients may be hepatitis B core antibody positive but must be surface antigen negative and without evidence of active infection.

Hepatitis C infection.

Pregnant or lactating. Patients of childbearing potential must use an effective method of contraception. The effects of chemotherapy, the subsequent transplant and the medications used after the transplant are highly likely to be harmful to a fetus. The effects upon breast milk are also unknown and may be harmful to the infant.

History of psychiatric disorder which may compromise compliance with transplant protocol, or which does not allow for appropriate informed consent (as determined by principal investigator or study chairman).

Exclusion Criteria Donor:

History of psychiatric disorder which may compromise compliance with transplant protocol, or which does not allow for appropriate informed consent.

History of hypertension that is not controlled by medication, stroke, or severe heart disease. Individuals with symptomatic angina will be considered to have severe heart disease will not be eligible to be a donor.

No other medical contraindications to stem cell donation (i.e. severe atherosclerosis, autoimmune disease, cerebrovascular accident, prior malignancy). Patients with a history of coronary artery bypass grafting or angioplasty will receive a cardiology evaluation and be considered on a case-by-case basis. Persons with a history of non-hematologic malignancy must have undergone potentially curative therapy for that malignancy and (1) have had no evidence of that disease for 5 years, and/or (2) be deemed at low risk for recurrence (less than or equal to 20% at 5 years). Such persons will be considered eligible for stem cell donation at the discretion of the principal investigator. Prospective donors with a history of non-hematologic malignancy who have received potentially curative therapy and are in remission, but whose estimated risk of recurrence is greater than 20% at 5 years, will be considered on an individual basis in consultation with the National Cancer Institute (NCI) Institutional Review Board (IRB).

Donors must not be pregnant. The effects of cytokine administration on a fetus are unknown. Donors of childbearing potential must use an effective method of contraception.

Anemia (Hb less than 11 gm/dl) or thrombocytopenia (platelets less than 100,000 per microliter).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2003-01-03 (Actual); Primary Completion 2014-09-25 (Actual); Study Completion 2014-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H Fowler, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Champlin RE. T-cell depletion for bone marrow transplantation: effects on graft rejection, graft-versus-host disease, graft-versus-leukemia, and survival. Cancer Treat Res. 1990;50:99-111. doi: 10.1007/978-1-4613-1493-6_6. PMID 1976361
- [Background] Giralt SA, Kolb HJ. Donor lymphocyte infusions. Curr Opin Oncol. 1996 Mar;8(2):96-102. doi: 10.1097/00001622-199603000-00004. PMID 8727301
- [Background] Martin PJ, Hansen JA, Torok-Storb B, Durnam D, Przepiorka D, O'Quigley J, Sanders J, Sullivan KM, Witherspoon RP, Deeg HJ, et al. Graft failure in patients receiving T cell-depleted HLA-identical allogeneic marrow transplants. Bone Marrow Transplant. 1988 Sep;3(5):445-56. PMID 3056552
- [Derived] Jamshed S, Fowler DH, Neelapu SS, Dean RM, Steinberg SM, Odom J, Bryant K, Hakim F, Bishop MR. EPOCH-F: a novel salvage regimen for multiple myeloma before reduced-intensity allogeneic hematopoietic SCT. Bone Marrow Transplant. 2011 May;46(5):676-81. doi: 10.1038/bmt.2010.173. Epub 2010 Jul 26. PMID 20661232
- [Derived] Baskar S, Suschak JM, Samija I, Srinivasan R, Childs RW, Pavletic SZ, Bishop MR, Rader C. A human monoclonal antibody drug and target discovery platform for B-cell chronic lymphocytic leukemia based on allogeneic hematopoietic stem cell transplantation and phage display. Blood. 2009 Nov 12;114(20):4494-502. doi: 10.1182/blood-2009-05-222786. Epub 2009 Aug 10. PMID 19667400

RESULTS

PARTICIPANT FLOW:
Groups:
- Recipient: Recipients will receive induction chemotherapy with fludarabine, cyclophosphamide, etoposide, doxorubicin, vincristine, and prednisone. (one cycle is 5 days on drug therapy followed by a 16 day rest period). Prior to the transplant procedure, recipients will receive conditioning therapy followed by the infusion of donor stem cells.
  Methotrexate: Recipients will receive 4 doses of methotrexate by vein after the transplant to help prevent graft-versus-host disease (GVHD).
  Cyclosporine: Recipients will receive cyclosporine by vein or by mouth for about 6 months after the transplant to help prevent graft-versus-host disease (GVHD).
Period: Overall Study
Arm/Group | Donor | Recipient
Started | 31 | 31
Completed | 19 | 17
Not Completed | 12 | 14
Not completed — Starting new study | 0 | 1
Not completed — Pt. to pursue treatment for progressive disease | 0 | 1
Not completed — Death of recipient | 8 | 8
Not completed — Recipient taken off study | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Donor | Recipient | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 27 | 52
  >=65 years | 6 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.98 (12.01) | 52.27 (12.33) | 52.12 (12.07)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 19 | 6 | 25
  Male | 11 | 23 | 34
  Missing | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 2
  White | 26 | 29 | 55
  Hispanic or Latino | 1 | 1 | 2
  Missing | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 31 | 31 | 62

OUTCOME MEASURES:

1. Primary Outcome: Number of Recipients Who Developed Grades I-IV Acute Graft Versus Host Disease (GVHD) Following a Combination of Cyclosporine and a Mini-dose Methotrexate Regimen for Graft Versus Host Disease (GVHD) Prophylaxis
Description: Here is the number of recipients who developed grades I-IV acute graft versus host disease (GVHD) following a combination of cyclosporine and a mini-dose methotrexate regimen for graft-versus-host disease (GVHD) prophylaxis. Grades I-IV acute GVHD clinical staging was assessed by the Glucksberg Criteria. Grade I-IV acute GVHD can occur in the skin, liver, and/or gut. Grade 1: rash < 25% body surface area (BSA), total bilirubin 2-3 mg/dl, and diarrhea 500-1000 ml/d. Grade 2: 25-50% BSA, total bilirubin 3-6 mg/dl, and diarrhea 1000-1500 ml/d. Grade 3: generalized erythroderma, total bilirubin 6-15 mg/dl, and diarrhea >1500 ml/d. Grade 4: desquamation and bullae, total bilirubin >15 mg/dl, and pain +/- ileus.
Time Frame: At least 100 days of follow-up post reduced-intensity stem cell transplantation (RIST)
Measure: Count of Participants; unit: Participants
Arm/Group | Recipient
Number analyzed (Participants) | 31
Participants
  Grade I GVHD | 1
  Grade II GVHD | 7
  Grade III GVHD | 6
  Grade IV GVHD | 0

2. Primary Outcome: Number of Recipients Who Developed Chronic Graft Versus Host Disease (GVHD) Following a Combination of Cyclosporine and a Mini-dose Methotrexate Regimen for Graft Versus Host Disease (GVHD) Prophylaxis
Description: Here is the number of recipients who developed chronic graft versus host disease (GVHD) following a combination of cyclosporine and a mini-dose methotrexate regimen for graft-versus-host disease (GVHD) prophylaxis. Grades I-IV chronic GVHD clinical staging was assessed by the Glucksberg Criteria. Grade I-IV chronic GVHD can occur in the skin, liver, and/or gut. Grade 1: rash < 25% body surface area (BSA), total bilirubin 2-3 mg/dl, and diarrhea 500-1000 ml/d. Grade 2: 25-50% BSA, total bilirubin 3-6 mg/dl, and diarrhea 1000-1500 ml/d. Grade 3: generalized erythroderma, total bilirubin 6-15 mg/dl, and diarrhea >1500 ml/d. Grade 4: desquamation and bullae, total bilirubin >15 mg/dl, and pain +/- ileus.
Time Frame: At least 100 days of follow-up post reduced-intensity stem cell transplantation (RIST)
Measure: Count of Participants; unit: Participants
Arm/Group | Recipient
Number analyzed (Participants) | 31
Participants | 23

3. Secondary Outcome: Percentage of Recipients Who Achieved Donor Chimerism at Day +14
Description: Recipients who achieved engraftment with donor chimerism. Engraftment is defined as a target peripheral blood cluster of differentiation 4 (CD4) count of 100 cells/ul after induction therapy.
Time Frame: Day+14
Measure: Number; unit: percentage of recipients
Arm/Group | Recipient
Number analyzed (Participants) | 31
percentage of recipients | 90

4. Secondary Outcome: Number of Recipients Evaluable Who Achieved Full Donor Chimerism at Day+100
Description: as for outcome 3
Time Frame: Day+100
Measure: Count of Participants; unit: Participants
Arm/Group | Recipient
Number analyzed (Participants) | 31
Participants | 29

5. Secondary Outcome: Median Cycles of Induction Chemotherapy With Fludarabine, Cyclophosphamide, Etoposide, Doxorubicin, Vincristine, and Prednisone Given to Recipients
Description: Median cycles of induction chemotherapy with fludarabine, cyclophosphamide, etoposide, doxorubicin, vincristine, and prednisone given to recipients.
Time Frame: Up to cycle 3
Measure: Median (Full Range); unit: Cycles
Arm/Group | Recipient
Number analyzed (Participants) | 31
Cycles | 2 [1 to 3]

6. Secondary Outcome: Median Time to Neutrophil Recovery
Description: Neutrophil recovery is defined as a neutrophil count ≥5000 µl for three consecutive days.
Time Frame: Up to 2 months after stem cell transplant
Population: The time to neutrophil recovery could not be determined precisely for 1 recipient who received granulocyte transfusions for an active infection following transplantation.
Measure: Median (Full Range); unit: Days
Arm/Group | Recipient
Number analyzed (Participants) | 30
Days | 14 [7 to 21]

7. Secondary Outcome: Median Time to Platelet Recovery
Description: Platelet recovery is defined as >50,000 mm3 platelet cell count after transfusion.
Time Frame: Up to 2 months after stem cell transplant
Population: Six recipients were not evaluable for platelet recovery > 20K because their platelet count never fell below that level (n=2) or because they were receiving aggressive platelet transfusions (n=4).
Measure: Median (Full Range); unit: Days
Arm/Group | Recipient
Number analyzed (Participants) | 25
Days | 13 [9 to 34]

8. Secondary Outcome: Number of Recipients With a Response to Reduced-intensity Stem Cell Transplantation (RIST)
Description: Complete remission (CR) is complete disappearance of all detectable signs and symptoms of lymphoma for a period of at least one month. Complete remission unconfirmed (CRu) is a residual lymph node mass > 1.5 cm in greatest transverse diameter will be considered CRu if it has regressed by more than 75% in the SPD, does not change over at least one month, is negative by PET or gallium, and is negative on any biopsies obtained (biopsy not required). Progressive disease (PD) is a 25% or greater increase in SPD of all measured lesions compared to the smallest previous measurements, or appearance of any new lesion(s).
Time Frame: At least 100 days after post reduced-intensity stem cell transplantation (RIST).
Measure: Count of Participants; unit: Participants
Arm/Group | Recipient
Number analyzed (Participants) | 31
Participants
  Complete Remission or Complete Remission Unconfirmed | 15
  Progressive Disease | 16

9. Other Pre Specified Outcome: Number of Recipients With Non-serious Adverse Events
Description: Here is the number of recipients with non-serious adverse events assessed by the Common Toxicity Criteria version 2.0. A non-serious adverse event is any untoward medical occurrence.
Time Frame: Date treatment consent signed to date off study, approximately 58 months and 13 days.
Population: Adverse events data were only collected for the recipients.
Measure: Count of Participants; unit: Participants
Arm/Group | Recipient
Number analyzed (Participants) | 31
Participants | 31

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 58 months and 13 days.
Description: Adverse events data were only collected for the recipients.
Arm/Group | Recipient
All-Cause Mortality (participants affected / at risk) | 11/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 31/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recipient (N=31)
Abdominal pain or cramping (Gastrointestinal disorders) | 8 (10)
Acute vascular leak syndrome (Vascular disorders) | 2 (2)
Alkaline phosphatase (Investigations) | 1 (2)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 2 (3)
Allergy-Other (Immune system disorders) | 4 (4)
Amylase (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 7 (9)
Arrhythmia - other (Cardiac disorders) | 1 (1)
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 1 (1)
Ascites (non-malignant) (Gastrointestinal disorders) | 2 (2)
Ataxia (incoordination) (Nervous system disorders) | 1 (1)
Autoimmune reaction (Immune system disorders) | 1 (1)
Bilirubin (Investigations) | 22 (47)
Bilirubin-graft versus host disease (GVHD) (Investigations) | 2 (3)
Bladder spasms (Renal and urinary disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Carbon monoxide diffusion capacity (DLCO) (Investigations) | 2 (2)
Cardiac left ventricular function (Cardiac disorders) | 3 (3)
Cataract (Eye disorders) | 1 (1)
Catheter-related infection (Infections and infestations) | 11 (15)
Chest pain (non-cardiac and non-pleuritic) (Musculoskeletal and connective tissue disorders) | 2 (2)
CNS hemorrhage/bleeding (Nervous system disorders) | 2 (2)
Cognitive disturbance/learning problems (Nervous system disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2)
Confusion (Psychiatric disorders) | 6 (7)
Conjunctivitis (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Constitutional symptoms - Other (General disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
CPK (creatine phosphokinase) (Investigations) | 2 (2)
Creatinine (Investigations) | 11 (15)
Diarrhea (without colostomy) (Gastrointestinal disorders) | 16 (27)
Diarrhea for BMT (Gastrointestinal disorders) | 9 (11)
DIC (disseminated intravascular coagulation) (Blood and lymphatic system disorders) | 1 (1)
Dry eye (Eye disorders) | 4 (4)
Dysphagia, esophagitis, odynophagia (painful swallowing) (Gastrointestinal disorders) | 3 (4)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dysuria (painful urination) (Renal and urinary disorders) | 4 (4)
Edema (General disorders) | 6 (7)
Endocrine-Other (Endocrine disorders) | 1 (1)
Erythema multiforme (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 6 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 21 (30) — (fever of unknown origin without clinically or microbiologically documented infection)
FEV1 (Investigations) | 4 (4)
Fever (in absence of neutropenia, where neutropenia is defined as AGC<1.0x109/L) (General disorders) | 24 (55)
Gastritis (Gastrointestinal disorders) | 2 (2)
GI-Other (Gastrointestinal disorders) | 3 (3)
Headache (Nervous system disorders) | 3 (6)
Hematuria (in the absence of vaginal bleeding) (Renal and urinary disorders) | 7 (7)
Hemoglobin (Hgb) (Investigations) | 28 (54)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia (Blood and lymphatic system disorders) | 5 (5)
Hemorrhage/bleeding without grade 3 or 4 thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Hepatic-Other (Hepatobiliary disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (12)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypertension (Vascular disorders) | 6 (7)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 (8)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 7 (11)
Hypotension (Vascular disorders) | 9 (11)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 12 (27)
Infection (documented clinically or microbiologically) with grade 3 or 4 neutropenia (Infections and infestations) | 22 (38)
Infection with unknown ANC (Infections and infestations) | 1 (1)
Infection without neutropenia (Infections and infestations) | 23 (86)
Infection, Other (Infections and infestations) | 14 (27)
Joint, muscle, or bone (osseous)-Other (Musculoskeletal and connective tissue disorders) | 2 (3)
Keratitis (corneal inflammation/corneal ulceration) (Eye disorders) | 1 (1)
Leukocytes (total WBC) (Investigations) | 1 (1)
Lymphatics (Blood and lymphatic system disorders) | 1 (1)
Melena/GI bleeding (Gastrointestinal disorders) | 1 (1)
Middle ear/hearing (Ear and labyrinth disorders) | 1 (1)
Mood alteration-depression (Psychiatric disorders) | 1 (1)
Mouth dryness (Gastrointestinal disorders) | 2 (2)
Mucositis due to radiation (Gastrointestinal disorders) | 2 (2)
Muscle weakness (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (muscle ache) (Musculoskeletal and connective tissue disorders) | 2 (2)
Myositis (inflammation/damage of muscle) (Infections and infestations) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (11)
Neurologic-Other (Nervous system disorders) | 2 (2)
Neuropathy motor (Nervous system disorders) | 2 (2)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 28 (58)
Neutrophils/granulocytes (ANC/AGC) for BMT (Investigations) | 31 (36)
Ocular-Other (Eye disorders) | 7 (7)
Pain-Other (General disorders) | 3 (3)
Platelets (Investigations) | 24 (49)
Platelets for BMT (Investigations) | 28 (33)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 8 (12)
Pericardial effusion/pericarditis (Cardiac disorders) | 3 (4)
Pulmonary-Other (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Radiation recall reaction (Injury, poisoning and procedural complications) | 1 (1) — (reaction following chemotherapy in the absence of additional radiation therapy
Rash/desquamation (Skin and subcutaneous tissue disorders) | 27 (49)
Rash-desquamation for BMT (Skin and subcutaneous tissue disorders) | 13 (19)
Renal/GU-Other (Renal and urinary disorders) | 2 (2)
Secondary Malignancy-Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Seizure(s) (Nervous system disorders) | 1 (1)
SGOT (AST) (Investigations) | 17 (36)
SGPT (ALT) (Investigations) | 18 (37)
Skin-Other (Skin and subcutaneous tissue disorders) | 3 (4)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Infections and infestations) | 9 (13)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) for BMT (Infections and infestations) | 7 (9)
Supraventricular arrhythmias (SVT/atrial fibrillation/flutter) (Cardiac disorders) | 5 (5)
Thrombosis/embolism (Vascular disorders) | 4 (6)
Transfusion: Platelets (Blood and lymphatic system disorders) | 2 (2)
Transfusion: pRBCs (Blood and lymphatic system disorders) | 5 (7)
Ureteral obstruction (Renal and urinary disorders) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 4 (4)
Ventricular arrhythmia (PVCs/bigeminy/trigeminy/ventricular tachycardia) (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Vision-blurred vision (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (9)
Weight gain (Investigations) | 6 (6)
Weight gain-veno-occlusive disease (VOD) (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2011-01-27): https://cdn.clinicaltrials.gov/large-docs/11/NCT00051311/Prot_SAP_000.pdf
  • Informed Consent Form: Donor Consent (2007-06-22): https://cdn.clinicaltrials.gov/large-docs/11/NCT00051311/ICF_001.pdf
  • Informed Consent Form: Recipient Consent (2004-07-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT00051311/ICF_002.pdf